CLINICAL TRIAL: NCT05528211
Title: Safety and Efficacy of Emergent Transcatheter Aortic Valve Implantation (TAVI) in Patients With Severe Aortic Valve Stenosis (AS): a Single-center, Prospective, Observational Cohort Study.
Brief Title: Safety and Efficacy of Emergent TAVI in Patients With Severe AS
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Chuanbao Li, Dr, Qilu Hospital of Shandong University
Other Study IDs: 20220823LCB
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation; Emergencies
MeSH Terms: conditions — Aortic Valve Stenosis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-centre, prospective, observational cohort study focusing on of patients suffering severe aortic valve stenosis (AS) undergoing emergent transcatheter aortic valve implantation (TAVI). AS patients undergoing emergent TAVI always have complicated clinical situations. Therefore, the aims of the study are to collect the incidence and outcomes of emergent TAVI in patients with severe symptomatic AS, to assess the safety and effectiveness of emergency TAVI system for severe AS, and to describe a more practical evidence of emergency TAVI system in severe AS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Every patient that diagnosed with severe aortic valve stenosis (evaluated by echocardiography: peak transaortic valve blood flow rate ≥4.0m/s, or mean transaortic valve pressure gradient ≥40mmHg (≥5.32kPa), or aortic Valve area <0.8cm2, or AVA<0.5cm2/m2);
2. Every patient that 1) required cardiopulmonary resuscitation due to cardiac arrest, or requiring external chest compressions during surgery (Salvage), 2) or has ongoing, refractory (difficult, complicated, and/or unmanageable) unrelenting cardiac compromise, with or without hemodynamic instability, and not responsive to any form of therapy except cardiac surgery (STS/ACC TVT defined "Urgent Status"), 3) or required urgent procedure during same hospitalization in order to minimize chance of further clinical deterioration (examples include, but are not limited to, worsening, sudden chest pain, heart failure, acute myocardial infarction, anatomy, intra-aortic balloon pump, unstable angina with intravenous nitroglycerin or rest angina) (STS/ACC TVT defined "Urgent Status");
3. Every patient that has been informed of the objectives of the study, agreed to participate, has signed the approved consent form, and was willing to accept all relevant examinations and clinical follow-up.

Exclusion Criteria:

1. Anatomically, the approach or aortic root is not suitable for transcatheter aortic valve implantation (TAVI).
2. Anatomical morphology or vascular diseases affecting the device approach.
3. Left ventricular outflow tract obstruction.
4. Primary dilated cardiomyopathy.
5. The echocardiogram indicates the presence of left ventricular thrombus.
6. Cannot tolerate anticoagulation and antiplatelet therapy.
7. Are allergic or resistant to nickel titanium alloys.
8. Active infective endocarditis, or other active infections affecting the effect of TAVI.
9. Severe disabling Alzheimer's disease.
10. Life expectancy< 6 months.
11. Other conditions (examples include poor compliance of patients and families) considered by the investigator to be inappropriate for participation in this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients with severe aortic valve stenosis undergoing emergency transcatheter aortic valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months post-TAVI
  including cardiac and non-cardiac deaths.

SECONDARY OUTCOMES:
The incidence of major adverse cardiovascular and cerebrovascular events (MACCEs) during the trial | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  Incidence of MACCEs (including mortality, disabling stroke, myocardial infarction, reoperation, arrhythmias and conduction blocks) during the trial.
Acute kidney injury | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  Incidence of acute kidney injury (kidney function was accessed by AKIN kidney function classification, including AKIN class II, AKIN class III and renal replacement therapy (RRT: hemodialysis, peritoneal dialysis, hemofiltration) ).
Permanent pacemaker implantation | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  Rate of patients implanted with permanent pacemaker.
Vascular complications (life-threatening or disabling) | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  including dissection, occlusion, rupture and bleeding of access vessels.
The incidence of other TAVI complications | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  including conversion to surgery, unexpected cardiopulmonary mechanical assistance, coronary artery occlusion, ventricular septal perforation, mitral valve injury or loss of function, pericardial tamponade, endocarditis, valve thrombosis, valve ectopic (displacement, embolization, misrelease), valve-in-valve, reoperation due to valve dysfunction, and so on.
Valve function | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  Doppler echocardiography was used to evaluate the valve performance at each follow-up point, including valve orifice area, mean aortic gradient, degree of valve regurgitation, moderate or above perivalvular leakage (PVL), and degree of aortic stenosis.
Cardiac function improvement | immediate, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-TAVI
  Doppler echocardiography was used to evaluate the heart function at each follow-up point, and cardiac function improvement is accessed by NYHA cardiac function classification, including NYHA class I, II, III and IV.
Device success rate | immediate post-TAVI
  Incidence of device success